CLINICAL TRIAL: NCT03342287
Title: Cognitive and Psychiatric Effects of Linaclotide on Patients With Irritable Bowel Syndrome-Constipation Predominant and Chronic Idiopathic Constipation
Brief Title: Cognitive and Psychiatric Effects of Linaclotide on Patients With Constipation
Status: Withdrawn | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Paul Moayyedi, Professor, McMaster University
Other Study IDs: 1088
Record Dates: First submitted 2016-03-01; First posted 2017-11-14 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Constipation; Irritable Bowel Syndrome
Keywords: gut microbiome; anxiety; depression; cognition
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and fecal samples collected.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaires — Questionnaires rating IBS symptoms, constipation, anxiety and depression
Other: cognitive evaluation — Administration of online cognitive battery
Other: Blood — Measurement of cytokines/inflammatory biomarkers
Other: Fecal sample — Measurement of the gut microbiome

SUMMARY:
Irritable Bowel syndrome - constipation predominant (IBS-C) is a chronic and disabling,disorder of the gut that is characterized by abdominal pain or discomfort. Approximately 50% of patients with IBS-C will also meet criteria for anxiety or depression.

Anti depressant medication is widely used in the treatment of IBS. Linaclotide is a novel medication for IBS that is also effective at relieving pain associated with IBS, which may be in part to signalling between the gut and the brain. However, the impact of Linaclotide on the psychiatric symptoms of anxiety and depression on IBS has not been investigated.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic, disabling functional gastrointestinal disorder that is characterized by abdominal pain or discomfort and a disturbance in bowel habit. It has long been recognized that psychological factors can be important in IBS, and that bi-directional signaling between the gut and the brain is likely involved in the pathophysiology of the syndrome. Approximately 50% of patients with IBS at a tertiary center will also meet criteria for anxiety or depression. Anti-depressant medications are widely used in the treatment of IBS, even without psychiatric comorbidity, with good evidence for both tricyclic antidepressants and selective serotonin reuptake inhibitors. Unfortunately both classes of anti-depressants have significant gastrointestinal side effects and a large number of patients cannot tolerate the medications.

Linaclotide, a guanylate cyclase agonist, has emerged as an important, novel treatment for patients with constipation-predominant IBS (IBS-C) and Chronic Idiopathic Constipation (CIC). Linaclotide is effective at relieving pain associated with IBS, which may be in part mediated by modulation of signaling between the gut and the brain. In this study the investigators will study the effect of Linaclotide on anxiety, depression and cognitive functioning in patients with IBS-C and CIC. If Linaclotide is also effective in treating anxiety and depression and improving cognitive functioning in patients with IBS-C and CIC, this will be an important therapeutic advance for the 50% of IBS patients with psychiatric comorbidity.

The investigators also propose to investigate the mechanisms by which Linaclotide may effect psychiatric symptoms and neuropsychological functioning by measuring changes in the gut microbiome and inflammatory biomarkers. The gut and the brain are intimately connected by several, bidirectional, signaling pathways including neural, humoral and immune mechanisms. The concept of the "gut-brain axis" has recently been supplanted by the "microbiota-gut-brain axis," emphasizing the important role the gut microbiota plays in mediating brain responses. The gut microbiota communicate with the brain through immune and neuronal pathways and some microbiota can directly secrete neurotransmitters such as serotonin, dopamine and gamma-aminobutyric acid (GABA) . In true bidirectional fashion, the brain can also influence the microbiota through the secretion of cortisol and sympathetic neurotransmission, changing gut motility, secretion and mucin production, which can affect the habitat of the resident microbiota and thereby alter the composition of the microbiota. Alterations in gut microbiota have been associated with irritable bowel syndrome in multiple studies.

Given the importance of the gut microbiota in mediating gut-brain responses, the investigators propose that the gut microbiota may play a direct role in the pathophysiology of anxiety and depression in patients with IBS. If Linaclotide is effective in reducing psychiatric and neuropsychological symptoms in patients with IBS, this may occur through changes in the gut microbiota, perhaps as a result of altered colonic motility and altered habitat of resident microbiota.

ELIGIBILITY:
Inclusion Criteria:

* IBS-C or CIC as defined by Rome III criteria
* able to provide and sign informed consent
* age 18-65 years

Exclusion Criteria:

* Previous diagnosis of bipolar, schizophrenia, or schizoaffective disorder
* psychosis
* active suicidal thoughts
* presence of a major neurocognitive disorder, delirium or other cognitive disorder
* active substance dependence ( including the use of cannabis more than 3 times per week
* active eating disorder
* pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBS-C or CIC starting on Linaclotide
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
To measure anxiety and depression using the Depression, Anxiety and Stress Scale (DASS) in patients with IBS-C and CIC before and after treatment with Linaclotide | Change from baseline to week 8

SECONDARY OUTCOMES:
To measure neuropsychological performance in Patients with IBS-C and CIC using a standardized neuropsychological assessment in patients (CNS vital signs) before and after treatment with Linaclotide | Change from baseline to week 8
  Neuropsychological testing will be performed using the standardized and validated CNS vital signs evaluation platform.
To determine changes in fecal microbiome profile before and after treatment with Linaclotide and whether these changes correlate with changes in psychiatric symptoms and cognition. | Change from baseline to week 8
  Fecal microbiome profile will be characterized using our in-house bioinformatics pipelines that provide measures of diversity between time points as well as differences in taxa between time points. Measurements will be aggregated to arrive at one reported value including diversity measures for microbiome analysis.
To determine changes in inflammatory biomarker profile before and after treatment with Linaclotide and whether these changes correlate with changes in psychiatric symptoms and cognition. | Change from baseline to week 8
  Inflammatory biomarkers measured will include IL-1, IL-6, TNF-alpha, IFN-gamma. Measurements will be aggregated to arrive at one reported value for average inflammatory biomarker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Moayyedi, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No